CLINICAL TRIAL: NCT01525420
Title: Improving Smoking Cessation Quitlines: Pilot Study of Acceptance Therapy
Acronym: TALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Consumer Wellness Solutions (Industry)
Responsible Party: Principal Investigator, Jonathan Bricker, Associate Member, Public Health Sciences, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7445
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): ACT: This is the experimental arm of the study. This included 5 weekly sessions of ACT therapy via telephone.
  Interventions: Behavioral: Acceptance Therapy (ACT)
- CBT (Active Comparator): CBT: This is the control arm of the study. This included 5 weekly sessions of CBT therapy via telephone.
  Interventions: Other: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Acceptance Therapy (ACT) — ACT
  Arms: ACT
Other: Cognitive Behavioral Therapy (CBT) — CBT
  Arms: CBT

SUMMARY:
The purpose of this study is to demonstrate that Acceptance Therapy (ACT's) implementation outcomes are at least as good as those of traditional cognitive behavioral therapy (CBT).

Implementation outcomes:

* end of treatment and 6-month follow-up data retention rates;
* intervention implementation quality;
* number & length of calls completed.

Comparison of each arm's implementation

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and older;
2. smokes at least 10 cigarettes daily and has done so for at least the past 12 months;
3. wants to quit smoking in the next 30 days;
4. willing to be randomly assigned to either group;
5. willing and able to speak and read in English;
6. willing and medically eligible to use nicotine replacement therapy (NRT),
7. currently resides in the U.S., and expects to continue for at least 12 months;
8. not participating in other smoking cessation interventions;
9. has regular access to a telephone.
10. has regular access to an email address.

Exclusion Criteria:

* The Exclusion criteria are the opposite of the Inclusion criteria listed above. In addition, the following exclusion criteria also apply:

  1. another member of household enrolled in the study;
  2. currently using medication or nicotine replacement products to help with quitting smoking;
  3. currently using any non-cigarette tobacco products;
  4. pregnant or breastfeeding;
  5. had a heart attack in last 30 days;
  6. within the last 6 months, diagnosed with angina, heart pain, or irregular heartbeat;
  7. serious adverse reactions to nicotine patches including anaphylaxis and related symptoms such as hives, respiratory difficulty, and/or angioedema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance & Commitment Therapy (ACT): ACT
  Acceptance & Commitment Therapy (ACT): ACT
  This is the experimental arm of the study. This included 5 weekly sessions of ACT therapy via telephone.
- Cognitive Behavioral Therapy (CBT): CBT
  Cognitive Behavioral Therapy (CBT): CBT
  This is the control arm of the study. This included 5 weekly sessions of CBT therapy via telephone.
Period: Overall Study
Arm/Group | Acceptance & Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Started | 59 | 62
Completed | 43 | 38
Not Completed | 16 | 24

BASELINE CHARACTERISTICS:
Groups:
- Acceptance & Commitment Therapy (ACT): ACT
  Acceptance & Commitment Therapy (ACT): This is the experimental arm of the study. This included 5 weekly sessions of ACT therapy via telephone.
- Cognitive Behavioral Therapy (CBT): CBT
  Cognitive Behavioral Therapy (CBT): ACT: This is the control arm of the study. This included 5 weekly sessions of CBT therapy via telephone.
- Total: Total of all reporting groups
Arm/Group | Acceptance & Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT) | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (9.5) | 38.6 (10.2) | 39.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 45 | 84
  Male | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Stopped Smoking by 6 Month Post Treatment
Description: 30-Day point prevalence abstinence at 6 months post treatment
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Acceptance & Commitment Therapy (ACT): ACT
  Acceptance & Commitment Therapy (ACT): ACT
Arm/Group | Acceptance & Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 59 | 62
participants | 18 | 14

2. Secondary Outcome: 7-day and 24-hour Point Prevalence Quit Rates
Description: 7-day and 24-hour point prevalence quit rates
Time Frame: 6-month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Acceptance & Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Serious Adverse Events (participants affected / at risk) | 2/59 | 0/62
Other Adverse Events (participants affected / at risk) | 0/59 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acceptance & Commitment Therapy (ACT) (N=59) | Cognitive Behavioral Therapy (CBT) (N=62)
No AE term known- see description (Social circumstances) | 1 | 0 — Unrelated to the study, bipolar participant hospitalized.
No AE term known - see description (Social circumstances) | 1 | 0 — Unrelated to the study, a participant was robbed and hospitalized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No